CLINICAL TRIAL: NCT02141139
Title: Suppression of Inflammation by Using NSAIDs During Peri-operative Period Can Affect the Prognosis of Breast Cancer.
Brief Title: Perioperative Inflammation and Breast Cancer Outcome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seok Jin Nam, Professor, Samsung Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-11-036
Record Dates: First submitted 2013-10-21; First posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Breast Neoplasms
Keywords: Anti-Inflammatory Agents, Non-Steroidal; Inflammation; Perioperative Period
MeSH Terms: conditions — Breast Neoplasms; Inflammation | interventions — Anti-Inflammatory Agents, Non-Steroidal; Ketorolac; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (No Intervention): no medication or acetaminophen
- NSAIDS (ketorolac intravenous, ibuprofen) (Experimental): ketorolac IV (just before surgery) and ibuprofen for 1 weeks
  Interventions: Drug: NSAIDS (ketorolac and ibuprofen)

INTERVENTIONS:
Drug: NSAIDS (ketorolac and ibuprofen)
  Arms: NSAIDS (ketorolac intravenous, ibuprofen)

SUMMARY:
It is increasingly recognized the NSAIDS (nonsteroidal antiinflammatory drug) might prevent the several cancers. In breast cancer, the role of NSAIDS (nonsteroidal antiinflammatory drug) has been suggested.However, there was no consistent results. surgery is main cause of inflammation for cancer patients. Therefore, we want to know the association between prevention of perioperative inflammation with NSAIDS and breast cancer outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who took the surgery

Exclusion Criteria:

* underlying medical disease (major heart disease, lung disease, coagulopathy)
* major psychologic disease (major depression, schizophrenia, manic disorder)
* pregnancy
* rheumatic disease patients

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1568 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 years

SECONDARY OUTCOMES:
overall survival | 5years

OTHER OUTCOMES:
neutrophil-lymphocyte ratio (NLR), albumin, inflammatory blood lab (CRP) | POD 1-2 weeks (immediate postoperative period)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea